CLINICAL TRIAL: NCT02956733
Title: Dermotaxis v/s Loop Suture Technique for Closure of Fasciotomy Wounds : a Study of 50 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Patiala (Other Government)
Responsible Party: Principal Investigator, Naveen Mittal, senior resident department of orthopaedics, Government Medical College, Patiala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/10/012461
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Inexpensive Closure of Fasciotomy Incisions Without the Need for Skin Grafting
Keywords: inexpensive, fasciotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dermotaxis (Active Comparator): In dermotaxis (Singhs skin traction) method two parallel kirschner wires (1.5mm) will be passed through the dermis on either side of the wound margins and interconnected by compression device consisting of threaded rod having two blocks and compression knob. Gradual compression will be applied daily at the rate of 1 turn/12hours on both sides of the wound.
  Interventions: Procedure: dermotaxis
- loop suture technique (Active Comparator): The loop suture technique involves using corrugated drains and Ethilon no.1. It is an extension of the purse string suture technique where a surgical suture is passed as a running stitch in and out along the edge of a wound in such a way that when the ends of the suture are drawn tight the wound is closed. Two corrugated drains (1 & 2) will be anchored to the skin adjacent to the fasciotomy incision using Ethilon no.1. Then the sutures will be passed from one edge of the wound through the skin and corrugated drain to the other in an alternating fashion.
  Interventions: Procedure: loop suture technique

INTERVENTIONS:
Procedure: dermotaxis — In dermotaxis (Singhs skin traction) method two parallel kirschner wires (1.5mm) will be passed through the dermis on either side of the wound margins and interconnected by compression device consisting of threaded rod having two blocks and compression knob. Gradual compression will be applied daily at the rate of 1 turn/12hours on both sides of the wound.
  Arms: dermotaxis
Procedure: loop suture technique — The loop suture technique involves using corrugated drains and Ethilon no.1. It is an extension of the purse string suture technique where a surgical suture is passed as a running stitch in and out along the edge of a wound in such a way that when the ends of the suture are drawn tight the wound is closed. Two corrugated drains (1 & 2) will be anchored to the skin adjacent to the fasciotomy incision using Ethilon no.1. Then the sutures will be passed from one edge of the wound through the skin and corrugated drain to the other in an alternating fashion.
  Arms: loop suture technique

SUMMARY:
The fasciotomy incisions lead to large, unsightly, chronic wounds after surgical intervention. The classic management was split thickness skin grafting but it leads to insensate skin with 23% of people upset by the appearance of the wound and 12% forced to changed occupation. Since no skin loss has occurred with the fasciotomy and utilizing the dermal properties of creep, stress relaxation and load cycling closure can be achieved in a better way. Our hypothesis is that using dermatotraction approximation could be done using inexpensive equipment readily available in any standard operating room.

DETAILED DESCRIPTION:
25 cases each of fasciotomy will be closed either by dermotaxis or loop suture technique with the inclusion criteria being closed fractures, no concomitant skin loss, fracture related compartment syndrome and fasciotomy within 36 hrs. The fasciotomy incision will be either closed in a single stage by loop suture technique or gradually by dermotaxis once the edema settled between 3-5 days. The results will be graded as excellent if approximation could be achieved, good if sutures have to be applied for protective care and poor if they have to be grafted. In dermotaxis (Singhs skin traction) method two parallel kirschner wires (1.5mm) will be passed through the dermis on either side of the wound margins and interconnected by compression device consisting of threaded rod having two blocks and compression knob. Gradual compression will be applied daily at the rate of 1 turn/12hours on both sides of the wound.

The loop suture technique involves using corrugated drains and Ethilon no.1. It is an extension of the purse string suture technique where a surgical suture is passed as a running stitch in and out along the edge of a wound in such a way that when the ends of the suture are drawn tight the wound is closed. Two corrugated drains (1 & 2) will be anchored to the skin adjacent to the fasciotomy incision using Ethilon no.1. Then the sutures will be passed from one edge of the wound through the skin and corrugated drain to the other in an alternating fashion.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria being closed fractures, no concomitant skin loss, fracture related compartment syndrome and fasciotomy within 36 hours.

Exclusion Criteria:

* The exclusion criteria was open fractures, skin loss, non-fracture related compartment syndrome and presentation after 36 hours

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
wound closure | 3 weeks
  The results will be graded as excellent if approximation could be achieved, good if sutures have to be applied for protective care and poor if they have to be grafted.

IPD SHARING:
Plan to Share IPD: Undecided